CLINICAL TRIAL: NCT05996536
Title: A Pilot Study to Assess Feasibility of Adipose Tissue Triglyceride (TG) Labelling in Familial Partial Lipodystrophy (FPLD)
Brief Title: Feasibility of Adipose Tissue Triglyceride (TG) Labelling in Familial Partial Lipodystrophy (FPLD)
Status: Recruiting | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10001651; 001651-DK
Record Dates: First submitted 2023-08-16; First posted 2023-08-18 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11-20

CONDITIONS: Lipodystrophy
Keywords: Lipodystrophy; Adipose Tissue
MeSH Terms: conditions — Lipodystrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-lipodystrophic controls: Non-lipodystrophic controls
- Partial Lipodystrophy: Partial Lipodystrophy

SUMMARY:
Background:

People with familial partial lipodystrophy (FPLD) do not store fat in the body normally. This can lead to serious illnesses such as diabetes and heart disease. To learn more about FPLD, researchers want to compare the fat tissue in people with this disease to the fat tissue of healthy people.

Objective:

To collect and analyze samples of fat tissue in people with and without FPLD.

Eligibility:

People aged 18 to 65 years with FPLD. Healthy adults are also needed.

Design:

Participants will be screened. They will have a physical exam. The size and shape of their body will be measured. They will have an imaging scan to measure their bones, muscle, and fat.

Participants will be given heavy water to drink at home. The water contains a tracer to help measure the fat in their blood. They will drink 1 vial 3 times a day.

After drinking the water for 9 days, participants will come to the clinic for a 3-day stay. They will eat only foods provided by the hospital; the foods will contain tracers. A needle will be inserted into a vein in the arm; participants will receive infusions of other tracers through this needle into their blood; this needle will also be used to draw blood samples for testing.

On their third day in the clinic, participants will have biopsies: Small samples of fat will be removed from under the skin on the belly and thigh.

Participants may return for a follow-up visit 8 days after leaving the clinic. Blood draws and fat tissue biopsies will be repeated.

DETAILED DESCRIPTION:
Study Description:

The feasibility of adipose tissue triglyceride labeling in patients with FPLD will be assessed in this non-interventional protocol. Specifically, subjects with FPLD (n=5) and control subjects without FPLD (n=5) will undergo isotope administration followed by abdominal and femoral subcutaneous fat biopsies.

Objectives:

Primary objective:

(1) To establish the technique of subcutaneous femoral adipose tissue biopsy in patients with FPLD, and subsequently, (2) to establish the feasibility of detecting labeled TG/FA in these adipose tissue biopsy samples.

Secondary objectives:

(1) To determine metabolic fluxes in healthy volunteers and patients with FPLD. (2) To determine if peripheral subcutaneous adipocytes are capable of fatty acid uptake and retention in patients with FPLD. (3) To assess standard metabolic parameters impacted by adipose fat storage capacity. (4) To assess different forms of circulating fat. (5) To determine feasibility of measuring adipose tissue lipoprotein lipase (LPL) activity.

Endpoints:

Primary Endpoints:

(1) Feasibility of performing subcutaneous femoral adipose tissue biopsy in patients with FPLD and (2) presence of detectable stable isotope labeling in adipose tissue specimens.

Secondary Endpoints:

(1) Blood labeling of glucose, glycerol, palmitate, and saponified fatty acids and other metabolites, as feasible; (2) quantity of stable isotope labeling in adipose tissue specimens; (3) blood glucose, insulin, NEFA, beta-OH-butyrate; (4) blood TG, VLDL, chylomicrons, NEFA and complete lipoprotein panel by NMR; (5) adipose tissue LPL activity and (6) adipose tissue histologic analysis.

ELIGIBILITY:
* INCLUSION CRITERIA:

Common inclusion criteria (FPLD and Controls):

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Stated willingness to comply with all study procedures and availability for the duration of the study
2. Age >= 18 and <= 65 years
3. Agreement to adhere to Lifestyle Considerations throughout study duration.
4. Weight stability (per the subject) within approximately 3 kg in the 3 months prior to screening, with no plans to actively gain or lose weight during the study period.

FPLD-specific inclusion criteria:

1. Clinical diagnosis of partial lipodystrophy based on reduction in adipose tissue outside the normal range in selected adipose depots (including, at a minimum, the gluteofemoral depot) with preservation of adipose tissue in other depots.
2. Adequate abdominal and thigh adipose tissue for feasible subcutaneous fat biopsy, as judged by the investigator.

CONTROL MATCHING CRITERIA:

When possible, control subjects will be individuals matched 1:1 with the FPLD subjects based on the following criteria (in order of priority). These criteria will be considered when assessing eligibility but are not strict inclusion criteria.

1. Sex
2. Age plus-minus 5 years
3. Diabetic status
4. Abdominal circumference plus-minus 10 cm
5. Height plus-minus 5 cm

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Uncontrolled diabetes, defined as HbA1C >8% at screening.
2. Use of insulin secretagogues (sulfonylureas) in week prior to Study Visit 1.
3. Changes in insulin dose >30% of total daily dose in the 2 weeks prior to Study Visit 1.
4. Use of niacin in the week prior to Study Visit 1.
5. Use of antiplatelets that cannot be safely held for the appropriate duration prior to each biopsy visit, including Plavix (one week prior to biopsy), aspirin (one week prior to biopsy) and NSAIDS (48 hours prior to biopsy).
6. Chronic use of anticoagulant medications that cannot be safely stopped for an appropriate duration of time prior to a biopsy procedure.
7. Lipemia defined as non-fasting triglycerides of >1000 mg/dL at screening.
8. Renal dysfunction defined as GFR <60 mL/min/1.73 m^2 at screening.
9. Consuming extreme macronutrient diet (e.g., very low-carbohydrate, high fat diets such as ketogenic, paleo or Atkins diets, among others).
10. Positive pregnancy test or breastfeeding at screening.
11. History of HIV, hepatitis B or C infection.
12. History of acquired lipodystrophy.
13. Clinically significant abnormalities in thyroid function, liver function, blood counts, or blood minerals as assessed by screening labs.
14. Inability to comply with planned study procedures.
15. Inability of subject to understand and the willingness to sign a written informed consent document.
16. Any condition which in the opinion of the investigator increases risk to subjects, prevents subject from complying with study procedures, prevents the subject from completing the study, or interferes with the interpretation of study results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with partial lipodystrophy and non-lipodystrophic controls.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of performing subcutaneous adipose tissue biopsy in patients with partial lipodystrophy. | 10 days
  Mass of adipose tissue obtained from each biopsy.
To determine the feasibility of detecting labeled TG/FA in femoral adipose tissue biopsy samples in patients with lipodystrophy, as compared to abdominal adipose tissue biopsy samples in the same patients, and as compared to controls. | 10 days
  Ability to detect labeled triglyceride and fatty acid in each biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca J Brown, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlies a publication will be shared.
Supporting Information: Study Protocol
Time Frame: Scientific data included in published manuscripts will be made available at the time of publication; all other generated scientific data will be shared no later than the termination date of the study.
Access Criteria: To maximize the appropriate sharing of scientific data and protect research participants privacy and confidentiality, reuse of this dataset should use the following Data Use Limitations (DULs) under Controlled Access that is made available by a data repository only after approval of the request by the repository's independent review panel process.@@@-Health/Medical/Biomedical - The dataset can only be used for studying health, medical, or biomedical conditions and does not include the study of population origins or ancestry.@@@-IRB Approval Required (IRB) - The requesting institution s IRB or equivalent body must approve the requested use.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001651-DK.html